CLINICAL TRIAL: NCT00375102
Title: Acupuncture and the Relaxation Response for Homeless Veterans With Substance Abuse
Brief Title: Acupuncture and the Relaxation Response for Substance Abuse
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: VA Boston Healthcare System (U.S. Federal Agency)
Collaborators: Samueli Institute for Information Biology (Other)
Responsible Party: Principal Investigator, Bei-Hung Chang, Health Research Scientist, VA Boston Healthcare System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1 EA-0000041
Record Dates: First submitted 2006-09-11; First posted 2006-09-12 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Substance Abuse
Keywords: acupuncture; relaxation response; homeless; veterans; randomized trials
MeSH Terms: conditions — Substance-Related Disorders | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Acup (Experimental): Acupuncture
  Interventions: Procedure: Acupuncture
- RR (Experimental): Relaxation Response
  Interventions: Behavioral: Relaxation Response
- UC (No Intervention): Usual Care

INTERVENTIONS:
Procedure: Acupuncture
  Arms: Acup
Behavioral: Relaxation Response
  Arms: RR

SUMMARY:
This one-year pilot study has two specific aims: 1. to determine the feasibility of conducting a randomized controlled trial of acupuncture and the relaxation response for substance abuse among homeless veterans who are in a domiciliary care program, and 2. to collect and analyze pilot data to estimate the effect size for planning a future larger study to fully test the hypothesis of the effectiveness of acupuncture and the RR in reducing cravings for substances (alcohol and drugs), and the corollary effects on quality of life.

DETAILED DESCRIPTION:
Substance abuse is one of the most important risk factors for homelessness. A high proportion of the US homeless population are veterans, in large part due to the high prevalence of substance abuse among veterans. Thus, effective substance abuse treatment in veterans is essential to preventing homelessness, as well as reintegrating those already homeless. Traditional substance abuse therapies have shown inconsistent effectiveness, suggesting a need for alternative therapies. Acupuncture and the relaxation response (RR) are two commonly used complementary and alternative medicine modalities that have shown benefit in some studies. However, they have not been studied in homeless veterans who have completed detoxification treatment and are in early remission. Acupuncture and the RR share common features, yet have distinct differences. Acupuncture has to be administered by acupuncturists, while RR elicitation is a self-care strategy that can be learned and practiced anytime and anywhere. We propose a pilot study to determine the feasibility of conducting a three-arm randomized controlled trial on veterans in the Bedford Domiciliary Care for Homeless Veterans program and to collect pilot data for planning future larger studies to test the effectiveness of acupuncture and the RR in reducing substance craving and improving anxiety and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Have a substance abuse or dependence problem of any type of substance
2. Stay in the domiciliary for at least 10 weeks after the study entry to complete the study.

Exclusion Criteria:

1. Schizophrenia or psychotic diagnoses
2. Bleeding disorders (hemophilia or thrombocytopenia)
3. An allergy to metals (needles).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2006-11; Primary Completion 2007-09 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Changes in self-reported substance craving rating from baseline to 10 week | baseline and 10 week follow up

SECONDARY OUTCOMES:
Changes in anxiety level from baseline to 10 week | baseline and 10 week follow up
Changes in quality of life from baseline to 10 week | baseline and 10 week follow up

CONTACTS AND LOCATIONS:
Overall Officials: Bei-Hung Chang, Sc.D., Principal Investigator — VA Boston Health Care System
Locations (1):
- Bedford VAMC, Bedford, Massachusetts, United States

REFERENCES:
- [Result] Chang BH, Sommers E. Acupuncture and relaxation response for craving and anxiety reduction among military veterans in recovery from substance use disorder. Am J Addict. 2014 Mar-Apr;23(2):129-36. doi: 10.1111/j.1521-0391.2013.12079.x. Epub 2013 Aug 30. PMID 25187049
- [Result] Chang BH, Elizabeth Sommers, Lawrence Herz, Acupuncture and relaxation response for substance use disorder recovery, Journal of Substance Use, 2010, 15(6): 390-401.